CLINICAL TRIAL: NCT04399876
Title: Pilot Study of an Implantable Microdevice for Evaluating Drug Responses in Situ in Prostate Cancer
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Oliver Jonas, Physician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-599; R01CA232174 (NIH)
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Radical Prostatectomy
Keywords: Prostate Cancer; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surgery Cohort (Experimental): Participant eligibility for intervention and selection of lesion for device placement
  - Surgery Cohort will undergo percutaneous placement of several microdevices in a selected tumor(s) prior to surgery. The microdevice in the surgery cohort will dwell in the tumor tissue for approximately 48 hours to allow time for tissue effects of the drugs in the microdevice reservoirs.
  Placement of at least 1, and up to 6, microdevices depending on the number of lesions, size and accessibility
  * Extirpative surgery will proceed according to standard-of-care procedures. The microdevice(s) will be removed surgically along with surrounding tumor tissue.
  * Standard of care treatment and follow-up of clinical course
  Interventions: Combination Product: Microdevice
- Ex-Vivo Cohort (Experimental): Each participant will undergo a screening process to determine their eligibility for microdevice placement, consisting of the following items:
  * Routine standard of care for radical prostatectomy.
  * Placement of implantable microdevice with multiple miniature drug reservoirs but no drug in prostate that have been removed
  * Ex vivo image guided removal using retrieval device
  * Standard of Care Treatment and follow-up of clinical course
  Interventions: Combination Product: Microdevice

INTERVENTIONS:
Combination Product: Microdevice — Surgery Cohort: Placement of 1-6 microdevices: Drugs chosen have all been FDA approved for the treatment of cancer (so therefore safe) and there are phase 2 or 3 data that the drug has efficacy in prostate cancer. Agents of interest included Abiraterone, Enzalutamide, Pembrolizumab, Ipilimumab, Carboplatin, Docetaxel, and Olaparib as well as combinations
  Ex vivo Cohort: Placement of multiple microdevices with miniature drug reservoirs but no drug is loaded into the removed prostate

SUMMARY:
In this research study, is assessing the feasibility of using an MR-guided implantable microdevice to measure tumor response to chemotherapy and other clinically relevant drugs in participants that have prostate cancer and are scheduled for a radical prostatectomy.

The name of the study intervention involved in this study is:

- Implantation of a MR-guided microdevice

DETAILED DESCRIPTION:
This research study is assessing the feasibility and safety of implanting and retrieving a 'microdevice' that releases up to 20 drugs directly within the prostate cancer lesion as a possible tool to evaluate the effectiveness of several approved cancer drugs against prostate cancer.

Participants will be identified with confirmed prostate cancer whose treatment plan includes surgery as a component of standard-of-care treatment.

The name of the study intervention involved in this study is:

* Implantation of a MR-guided microdevice .
* It is expected that about 35 people will take part in this research study; 5 in the Ex Vivo Cohort and 30 in Surgery Cohort.

  * Ex Vivo Cohort will undergo placement of microdevice in the prostate after its surgical removal.
  * Surgery Cohort will undergo percutaneous placement of several microdevices in a selected tumor prior to surgery.

This research study is a Pilot Study, which is the first-time investigators are examining this study intervention. The FDA (the U.S. Food and Drug Administration) has not approved the implantation of the microdevice for this specific disease, but usage of this has been approved for other uses.

ELIGIBILITY:
Eligibility Criteria: Ex Vivo Cohort

* Inclusion Criteria

  * Participants must have the ability to understand and the willingness to sign a written informed consent document.
  * Planned radical prostatectomy for prostate cancer.
  * Participants must be 22 years of age or older.
* Exclusion Criteria -- Unwillingness to sign informed consent.

Eligibility Criteria: Surgical Cohort

* Inclusion Criteria

  * Participants must have the ability to understand and the willingness to sign a written informed consent document.
  * Patients must have the ability to understand and the willingness to sign a written informed consent document at the study site when both the investigator and participant are at the same location, or remotely (e.g., at the participant's home or another convenient venue) where the participant reviews the consent document with the Licensed Physician Investigator over secure Zoom. The electronic consent system, Adobe, ensures the participant electronically signing the informed consent is the subject who will be participating in the research study.
  * Participants must present with prostate cancer falling into an intermediate or high risk category to include features: Gleason score 3+4 or higher, greater than 3 biopsy cores positive and ≥50% of 1 core positive for carcinoma, and an MRI-visible lesion concerning for PCa in the region of the positive biopsy.
  * Participants must be 22 years of age or older.
  * Participants must be evaluated by a urologic oncologist who will determine the clinically appropriate treatment strategy based on clinical history and extent of disease.
  * Participants must be deemed medically stable to undergo both percutaneous procedures and standard-of-care surgical procedures by their treating surgeon.
  * Participants must have undergone multi-parametric prostate MRI that both assesses the extent of disease and allows the research team to assess for study eligibility. This will have been done as part of the standard-of-care. Abnormal imaging will be correlated with the biopsy findings to maximize the likelihood of the device being put in the lesion. If the images are not adequate, the MRI scan will be repeated at BWH/DFCI, again as part of standard-of-care management.
  * The participant's case must be reviewed by representatives of urologic oncology and interventional radiology to assess the following factors:

    * Participant is clinically stable to undergo biopsy procedure(s) and surgical procedures.
    * Participant has sufficient volume of disease as shown by MRI to allow implantation of the microdevice.
    * A lesion can be selected where the microdevice is to be implanted that is a) amenable to percutaneous placement, and b) amenable to removal at the time of primary surgery
  * Participants must be willing to undergo research-related genetic sequencing (somatic and germline) and data management, including the deposition of de-identified genetic sequencing data in NIH central data repositories.
  * For men: agreement to refrain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm during the treatment period and for 28 days after the last dose of ipatasertib.
* Exclusion Criteria

  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit the safety of a biopsy and/or surgery.
  * Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or biopsy procedures.

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as defined in the CTCAE v4.0 | From the time of arrival to interventional radiology for microdevice placement up to 6 weeks.
  Safety of microdevice placement and removal based on assessment of adverse events
Number of Participants with successful surgical Placement and retrieval of Microdevice | 48 Hours
  * Feasibility of microdevice placement based on the ability in the Surgical Cohort to percutaneously place and surgically retrieve the device with sufficient tissue, of sufficient quality, for downstream histopathology analysis and interpretation.
  * In the Surgical Cohort, if not more than 1 IMD per patient fails to be percutaneously placed and surgically retrieved with sufficient tissue of sufficient quality for downstream histopathology analysis and interpretation, we would consider this procedure to be a success. If at least 23/30 Surgical Cohort patients have successful procedures, as previously defined, we would consider this approach feasible. The 90% CI for 23 out of 30 successes is (60.6%, 88.5%) and thus excluding a 60% success rate which is considered as too low.

SECONDARY OUTCOMES:
Local intratumor response | 48 Hours
  measure local intratumor response to clinically relevant cytotoxic agents and small molecule drugs in prostate cancers using quantitative histopathologic assessment of tumor tissue.
  All inferences of secondary endpoints will use two-sided alpha = 0.05 and report 95% confidence intervals with any point estimates. Descriptive statistics will be used to summarize the quantitative measurements of apoptosis, proliferation, DNA repair, etc. for drug-treated regions compared to vehicle-treated regions. At least two separate regions will contain vehicle to account for tumor heterogeneity.
Intratumor heterogeneity in drug response | 48 Hours
  comparing the extent of tumor response to drug among different locations in a single tumor with multiple microdevice.
  All inferences of secondary endpoints will use two-sided alpha = 0.05 and report 95% confidence intervals with any point estimates.
Biomarkers of drug response | 48 Hours
  immune infiltrates, in the local tumor tissue adjacent to the microdevice, and to perform a preliminary assessment of the correlation between these features and extent of tumor response with the microdevice All inferences of secondary endpoints will use two-sided alpha = 0.05 and report 95% confidence intervals with any point estimates.
Genetic features of the tumor tissue | 48 Hours
  To determine the genetic features of the tumor tissue adjacent to the microdevice (e.g. whole exome sequencing, whole transcriptome sequencing) and to perform a preliminary assessment of the correlation between known genetic markers of drug sensitivity or resistance and extent of tumor response with the microdevice Genetic alterations will be catalogued in terms of single nucleotide variants, insertions/deletions, and copy number changes and will be primarily reported in a descriptive manner. Preliminary correlations between a specific genetic feature and specific clinical features will be tested using the Chi-squared/Fisher's exact test for categorical variables or the T-test or Wilcoxon Rank-Sum test for continuous variables

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Kibel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Stone BV, Dominas CA, Bhagavatula SK, Ahn SW, Tatarova Z, Jakubik J, Matthew D, Mossanen M, Furtado D, Tuncali K, Hirsch MS, Hata N, Tempany C, Jonas O, Kibel AS. Novel Intraprostatic Magnetic Resonance-Guided Implantation of Multidrug-Eluting Microdevice for Testing of Systemic Therapy Agents In Situ: Proof of Concept in Intermediate-Risk and High-Risk Prostate Cancer. J Urol. 2025 Feb;213(2):173-182. doi: 10.1097/JU.0000000000004269. Epub 2024 Sep 30. PMID 39348711